CLINICAL TRIAL: NCT06510634
Title: Effectiveness and Safety of Endovascular Treatment vs. Best Medical Treatment in Patients With Vertebrobasilar Artery Occlusion Presenting Beyond 24 Hours of Last Known Well：a Prospective, Multicenter Registry Study
Brief Title: Triage of Patients Presenting Beyond 24 Hours With Ischemic Stroke Due to Vertebrobasilar Artery Occlusion
Acronym: VBAO-LATE
Status: Enrolling by invitation | Type: Observational
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Ming Wei, Chief Physician, Tianjin Huanhu Hospital
Other Study IDs: TJHH-2024-WM51
Record Dates: First submitted 2024-07-14; First posted 2024-07-19 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- endovascular thrombectomy group: The EVT group would include Stent retriever thrombectomy; Aspiration; Balloon angioplasty and/or stenting; Intra-arterial medication; Combination
  Interventions: Other: Endovascular Therapy
- best medical treatment gruop: BMM consisted of IVT antiplatelet drugs, anticoagulation, or combinations of these treatment modalities according to institutional guidelines.
  Interventions: Other: Endovascular Therapy

INTERVENTIONS:
Other: Endovascular Therapy — Endovascular therapy, as an adjunct to standard stroke therapy, may be beneficial for a very select population of patients who present with an acute ischemic stroke and have a proven large, proximal occlusion on imaging.
  Endovascular therapy includes any one or more of the following:
  Intra-arterial thrombolytic therapy, aspiration, stent retrieval, or a combination of multiple mechanical devices.

SUMMARY:
Endovascular thrombectomy (EVT) for posterior circulation occlusion is generally performed within a window of less than 24 hours from the time the patient was last known well (LKW). The efficacy and safety of EVT beyond the 24-hour window remain uncertain.

ELIGIBILITY:
Inclusion Criteria:

1. age≥18 years.;
2. blockage in the vertebrobasilar artery, including the vertebral artery or basilar artery, determined using computed tomographic angiography (CTA)/ magnetic resonance angiography (MRA)/digital subtraction angiography (DSA);
3. VBAO occurrence more than 24 hours from LKW;
4. none to mild premorbid disability defined by modified Rankin Scale (mRS) score ≤2;
5. informed consent before enrollment in the clinical trials.

Exclusion Criteria:

1. neuroimaging evidence of cerebral hemorrhage on presentation;
2. lack of follow up information on outcomes at 90 days
3. serious, advanced, or terminal illness.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study is a prospective, multicenter cohort study, which analyzed the prospectively databases of 11 stroke centers.Including patients with ischemic stroke due to vertebrobasilar artery beyond 24 hours from last known well.
Sampling Method: Non-Probability Sample
Enrollment: 236 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
proportion of patients with Modified ranking scale (mRS) (0-3) at 90 days | 90(±14)days
  A 0-6 scale running from perfect health without symptoms to death.

SECONDARY OUTCOMES:
distribution of patients with Modified ranking scale (mRS) (0-3) at 90 days | 90(±14)days
  A 0-6 scale running from perfect health without symptoms to death.
Mortality within 90 days | 90(±14)days
  mortality of any causes.
Incidence of symptomatic intracranial haemorrhage | 90(±14)days
  Symptomatic intracranial hemorrhage was characterized as any type of intracranial hemorrhage observed on follow-up imaging between 22 and 36 hours and 7 days after stroke onset, accompanied by an increase of at least 4 points on the NIHSS from baseline or the lowest value within 7 days, or resulting in mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided